CLINICAL TRIAL: NCT06087185
Title: Evaluation of the Effect of Mindful Eating in Patients With Anxiety and Obesity.
Brief Title: Obesity and Mindful Eating in Patients With Anxiety
Acronym: OMETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 66476322.5.0000.5327; 2022-0551 (Other: HCPA)
Record Dates: First submitted 2023-08-29; First posted 2023-10-17 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Obesity; Eating Behavior; Mindfulness; Inflammation; Self-Control
Keywords: Anxiety; Obesity; Eating Behavior; Mindfulness
MeSH Terms: conditions — Anxiety Disorders; Obesity; Feeding Behavior; Inflammation; Self-Control | interventions — Mindfulness; Eating

STUDY DESIGN:
Intervention Model Description: This is a Randomized Clinical Trial (RCT) comparing the effectiveness of the adapted Mindful Eating protocol to the control with exposure to videos promoting quality of life in adults with anxiety and obesity.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindful Eating Group (Experimental): Mindful Eating practices will be taught during a weekly meeting lasting 150 minutes and individuals will be encouraged to integrate the practices learned into their daily lives, for at least 15 minutes a day, being progressively integrated into the other practices that will be taught in subsequent weeks. There will be a WhatsApp group with reminders during the week and audio for guided practice.
  Interventions: Behavioral: Mindful Eating
- Video Group (Active Comparator): Composed of 5 videos sent weekly produced by trained professionals. The topics discussed will be relevant to the management of anxiety in general and lifestyle changes.
  Video 1: Psychoeducation of anxiety. Video 2: Healthy eating. Video 3: Sleep hygiene. Video 4: Physical activity. Video 5: Substance use. This protocol used as a control was effective as a Psychoeducation Group in improving anxiety symptoms in patients with generalized anxiety disorder.
  Interventions: Behavioral: Video Group

INTERVENTIONS:
Behavioral: Mindful Eating — Mindful Eating practices will be taught during a weekly meeting lasting 150 minutes and individuals will be encouraged to integrate the practices learned into their daily lives, for at least 15 minutes a day, being progressively integrated into the other practices that will be taught in subsequent weeks. There will be a WhatsApp group with reminders during the week and audio for guided practice.
  Other Names: Mindfulness; Eat for Life protocol
  Arms: Mindful Eating Group
Behavioral: Video Group — Composed of 5 videos sent weekly produced by trained professionals. The topics discussed will be relevant to the management of anxiety in general and lifestyle changes.
  Video 1: Psychoeducation of anxiety. Video 2: Healthy eating. Video 3: Sleep hygiene. Video 4: Physical activity. Video 5: Substance use. This protocol used as a control was effective as a Psychoeducation Group in improving anxiety symptoms in patients with generalized anxiety disorder.
  Arms: Video Group

SUMMARY:
Background: Obesity is chronic disease with high prevalence rates, functional disability and difficult long-term management. Anxiety is one of the most common psychological disorders in obesity, and when associated with other factors such as emotional eating and emotional dysregulation, it impairs treatment and interferes with lifestyle changes. Finding an intervention that improves the eating behavior of these patients and facilitates adherence to obesity treatment, associated with less emotional distress, is of great clinical interest. Objective: The aim of this study is to evaluate the effectiveness of the Mindful Eating (ME) intervention on neurocognitive and behavioral outcomes in patients with obesity and anxiety compared to the control group with exposure to videos promoting quality of life. Methods: A five-weeks randomized clinical trial will be performed with 52 patients in adulthood. The Mindful Eating intervention group will receive an online protocol with one meeting per week. This is a protocol that has been adapted for five weeks and consists of a group intervention with 10-15 participants. Mindfulness, Mindful Eating and Self-Compassion training will be based on the Eat for Life protocol. The control group will receive five videos of psychoeducation, one topic per week. After, all participants will receive lifestyle advices, a first-line "treatment-as-usual" to obesity. There will be a face-to-face assessment with anthropometric, behavioral and biological measurements pre and post-intervention. The outcomes may help in understanding the mechanisms underlying the change in eating behavior, in order to direct new therapeutic strategies for the treatment of anxiety and obesity comorbidities.

DETAILED DESCRIPTION:
This study is the second phase of a cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 50 years old;
* Inclusion for Generalized Anxiety Disorder (GAD):

Primary GAD diagnosed by the M.I.N.I.;

✔Inclusion for Obesity: Obesity BMI grade I (between 30.0 and 34.9); Obesity BMI grade II (between 35.0 and 39.9)

Exclusion Criteria:

* In individuals with obesity or control only, not having any psychiatric disorder;
* In individuals with only GAD or control, do not have a BMI above 25.
* In individuals with GAD, not having a diagnosis of primary or severe depression;
* Being under psychopharmacological, psychotherapeutic or nutritional treatment;
* Bipolar Disorder, Psychotic Disorder, Substance Use Disorder (except Tobacco) in the last 6 months or Suicidal Ideation in the last 6 months (M.I.N.I);
* Have a clinical instability or immobility;
* Being in Pregnancy or Lactation;
* Antisocial Personality Disorder;
* Eating Disorder.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Inhibitory Control | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in the performance in Go/No-go task compared to the control group with exposure to videos. This paradigm consists of the presentation of neutral images and food images on a computer screen (presented randomly, with a millisecond interval between them) and the participant must press or not press a key according to the researcher's instructions. The participant will be instructed to press the specific "Go" key when certain neutral images are viewed (office objects and bathroom objects). When food images and another class of neutral images (sports objects) are viewed, the participant will be instructed not to press any key and just wait (No Go). The "Go/No Go" paradigm, which has high reliability and replicability, makes it possible to evaluate inhibitory control, considering the commissioned number of errors in the No Go outcome.

SECONDARY OUTCOMES:
Change in Inflammatory Markers | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Protein C-reactive and Interleukine-6 compared to the control group with exposure to videos.
Change in Emotional Regulation | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Difficulties in Emotion Regulation Scale (DERS) compared to the control group with exposure to videos. It is an instrument that assesses levels of emotional dysregulation in six domains. Contains 36 items on a 5-point Likert scale from 1 to 5.
Change in Self-Compassion | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Self-Compassion Scale (SCS) compared to the control group with exposure to videos. The self-compassion scale was designed to measure self-compassion in three components: self-judgment versus self-kindness (SJ-SK), sense of isolation versus common humanity (I-CH), over-identification versus mindfulness (OI-M). Respondents must rate how they usually behave in difficult times, according to a scale with 26 5-point items. Therefore, the higher the total SCS score, the more self-compassionate the individual.
Change in Impulsivity | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Barratt Impulsiveness Scale (BIS-11) compared to the control group with exposure to videos. The self-report scale developed by Barratt to assess these dimensions of impulsivity is composed of 20 questions for Inhibitory Control and 8 for Lack of Planning. The higher the score, the greater the level of impulsiveness.
Change in Emotional Eating | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Factor Eating Questionnaire (TFEQ-R21) compared to the control group with exposure to videos. This questionnaire is a self-administered instrument that assesses cognitive restriction behaviors (six questions), emotional eating (six questions) and uncontrolled eating (nine questions) and has good internal consistency. It has a total of 21 questions in which individuals rate the statement as true or false on a four-point scale, with "1" being completely true and "4" being completely false.
Change in Binge Eating | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Binge Eating Scale (BES) compared to the control group with exposure to videos. The BES is a self-administered Likert questionnaire, consisting of a list of 16 items and 62 statements, from which the one that best represents the individual's response must be selected for each item. Each statement corresponds to a number of points from 0 to 3, ranging from absence ("0") to maximum severity ("3") of binge eating.
Change in Body Appreciation | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Body Appreciation Scale (BAS) compared to the control group with exposure to videos. The BAS is a 13-item questionnaire designed to assess the degree of body appreciation. Items are rated on a five-point scale ranging from one (never) to five (always). Higher scores reflect greater body appreciation.
Change in Parental Bonding | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of The Parental Bonding Instrument (PBI) compared to the control group with exposure to videos.It is used to measure parental behavior as perceived by the offspring. The instrument consists of 25 items: 12 'care' items and 13 'protection' items. Raters are asked to rate the parents' behavior as they remember it in the first 16 years of their lives. For mothers, the cut-off point between the high and low scores is 27.0 and for the protection score it is 13.5. For parents, a care score of 24.0 and a protection score of 12.5.
Change in Early Memories | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Early Memories of Warmth and Safeness Scale (EMWSS) compared to the control group with exposure to videos. The EMWSS is a measure that assesses emotional memories of being protected, loved and cared for by adults. The scale assesses recall of positive feelings particularly of safety, warmth and care during childhood. It is a 21-item Likert-type scale (from 0=never to 4=Yes, most of the time).
Change in Early Life Experiences | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of The Early Life Experiences Scale (ELES) compared to the control group with exposure to videos. This scale was designed to measure recall of perceived threat and subordination in childhood. The scale, therefore, is composed of 15 items focused on recalling the perceived threat (six items) and feeling subordinate and acting submissively (nine items). The response measure consists of a Likert-type scale assessing how often and how true each statement was for them in their childhood.
Change in Experiences in Close Relationships | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Experiences in Close Relationships - Relationship Structures Questionnaire (ECR-RS) compared to the control group with exposure to videos. The ECR-RS evaluates the bonding styles established in relationships with close people: father, mother, partner and friend. Each relationship is rated on a scale that theoretically comprises two factors: anxious and avoidant attachment. The total score for each subscale is the average of the items and ranges from 1 to 7, with higher scores indicating greater avoidant or anxious attachment.
Change in Weight Bias Internalization | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Weight Bias Internalization Scale (WBIS) compared to the control group with exposure to videos. The scale score ranges from 11 to 77 points, with items 1 and 9 evaluated with reverse scoring. The WBIS is self-administered and has no cutoff point, however, higher scores indicate greater internalization of weight stigma.
Change in BMI | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of Body Mass Index (BMI) compared to the control group with exposure to videos.
Change in Body Fat - Bioimpedance index | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of body fat percentage compared to the control group with exposure to videos.
Change in Insulin resistance | 5 weeks
  To evaluate the effectiveness of the Mindful Eating (ME) intervention in levels of HOMA index compared to the control group with exposure to videos. The Homeostasis Model Assessment (HOMA) estimates steady state beta cell function and insulin sensitivity, as percentages of a normal reference population.

CONTACTS AND LOCATIONS:
Overall Officials: Gisele G Manfro, PhD, Study Director — Federal University of Health Science of Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: OMETA Instagram — https://instagram.com/ometaprojeto?igshid=MzRlODBiNWFlZA==